CLINICAL TRIAL: NCT02661061
Title: Ketamine for Relapse Prevention in Recurrent Depressive Disorder: a Randomised, Controlled, Pilot Trial: the KINDRED Trial
Brief Title: Ketamine for Relapse Prevention in Recurrent Depressive Disorder
Acronym: KINDRED
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: St Patrick's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Prof Declan McLoughlin, Professor, St Patrick's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20/15; 2015-002020-37 (EudraCT Number)
Record Dates: First submitted 2015-12-10; First posted 2016-01-22 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Depression; Relapse; Recurrent Depressive Disorder; Major Depressive Disorder
Keywords: ketamine; glutamate; relapse prevention
MeSH Terms: conditions — Depression; Recurrence; Depressive Disorder; Depressive Disorder, Major | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: A randomised, double-blind, placebo-controlled study designed to assess feasibility of recruitment, randomisation and retention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking took place by sealed envelope random allocation and double blinding of participants and raters was assessed throughout. The anaesthesiologist administering infusions was aware of the allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Trial Interventions: participants will receive four two-weekly infusions of ketamine at 0.05mg/kg. All infusions will be administered by a consultant anaesthetist.
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Trial Interventions: participants will receive four two-weekly infusions of midazolam at 0.045mg/kg. All infusions will be administered by a consultant anaesthetist.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — A sub-anaesthetic dose of ketamine will be administered in four infusions, each two weeks apart.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Midazolam — A sub-anaesthetic dose of midazolam will be administered in four infusions, each two weeks apart.
  Other Names: Hypnovel
  Arms: Midazolam

SUMMARY:
Randomised, controlled, parallel-group, pilot clinical trial of ketamine vs. midazolam for depression relapse prevention in persons at high risk. The main purpose of the pilot study is to assess trial processes to help inform a future definitive trial.

DETAILED DESCRIPTION:
Participants will be recruited at admission to St Patrick's University Hospital for treatment of the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV)-diagnosed recurrent unipolar depression and followed-up weekly to assess recovery according to standard criteria. Blood samples for epigenetic studies will be taken at baseline. Treatment-as-usual will continue throughout the entire trial. Participants who meet standardised response criteria will then be invited to be randomised to course of four two-weekly ketamine or midazolam (active comparator) infusions. Block randomisation will be independently performed. Physical, psychotomimetic and cognitive outcomes will be monitored before, during and after infusions. Blood samples will be taken at four time-points in the first infusion session and before the final infusion for neuroplasticity biomarker studies.Trial Interventions: participants will receive four two-weekly infusions of either ketamine at 0.05mg/kg or midazolam at 0.045mg/kg. All infusions will be administered by a consultant anaesthetist. Repeated infusions of ketamine have been shown to be safe and well-tolerated by patients with mental illness. Minor haemodynamic changes and psychotomimetic side-effects can occur and will be assessed regularly during infusions and for 200 minutes afterwards.

Participants will be followed up over six months to assess for relapse according to standardised criteria. This is the highest-risk period for relapse and investigators hypothesize that ketamine will provide additional neurotrophic support (assessed by the laboratory biomarker project) which will result in lower relapse rates when compared to midazolam.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Hamilton Rating Scale for Depression, 24-item (HRSD-24) score of ≥21
* Voluntary admission for treatment of acute depressive episode
* Meet DSM-IV criteria for recurrent depressive disorder (RDD): ≥2 previous depressive episodes with at least 2-months(consecutive) subthreshold or no symptoms in between PLUS(to enrich the sample for those at high risk for relapse) must also have experienced ≥3 major depressive episodes(including index episode) within the previous 2 years

For the randomised pilot trial, RDD patients must have:

* received antidepressant treatment for the acute depressive episode(pharmacological, psychotherapeutic or multidisciplinary)
* ≥60% decrease from baseline HRSD-24 score and score ≤16
* Standardised Mini-Mental State Examination (sMMSE) score of ≥24
* able to provide informed consent

Exclusion Criteria:

* Current involuntary admission
* Medical condition rendering unfit for ketamine/midazolam
* Active suicidal intention
* Dementia
* History of Axis 1 diagnosis other than RDD
* Electroconvulsive therapy (ECT) for treatment of current depressive episode
* Alcohol/substance abuse in previous six months
* Pregnancy or inability to confirm use of adequate contraception during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-12; Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Declan McLoughlin, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- St Patrick's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
None envisaged: data will be anonymised

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were inpatients at St Patrick's Mental Health Services admitted for treatment of an acute depressive episode with a previous history of depression
Pre-assignment Details: Participants were randomised from n=28 participants in an observational phase, all of whom were receiving inpatient treatment for recurrent depressive disorder. Participants were monitored weekly for response to treatment and those who responded were invited to be randomised.
Period: Overall Study
Arm/Group | Ketamine | Midazolam
Started | 5 | 4
Completed | 3 | 2
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Midazolam | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate for Randomised Treatment Phase
Description: The outcomes for this pilot trial are process outcomes, primarily rates of recruitment and retention. Thus, the completion rate for the randomised treatment phase is the primary outcome. The study is not designed to assess efficacy.
Time Frame: 2 years
Population: All randomised participants who received one infusion were analysed (intention to treat)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 5 | 4
Participants | 3 | 2

2. Secondary Outcome: Depression Relapse Rate During Treatment and Follow-up Phase
Description: Clinical outcomes are secondary in this pilot trial. The 24-item Hamilton Rating Scale for Depression (HRSD-24) was used to assess for the main clinical outcome, the relapse rate over six months. Criteria for relapse are ≥10 point increase in HRSD-24 compared to baseline score plus HRSD ≥16; in addition, increase in the HRSD should be maintained one week later (if indicated, additional follow-ups will be arranged). Hospital admission, and deliberate self-harm/suicide also constitute relapse. Relapse may also occur during the eight-week treatment phase and is captured here.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 5 | 4
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse event information was collected over the entire study time frame, 29 months, from December 2015 to May 2018. Individual participants were assessed over an approximately seven-month period including their inpatient admission, eight-week randomised treatment phase, and 26-week follow-up period.
Description: Tolerability of the trial agents was assessed at multiple points before, during and after treatment sessions using a battery of assessments used in assessing for physical and psychotomimetic side effects of ketamine (CADSS, BPRS, PRISE and YMRS), standard in the field of ketamine clinical trials for depression, as well as assessment of physical health parameters before, during and after assessments.
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=5) | Midazolam (N=4)
Delayed hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0) — Possible delayed hypersensitivity reaction a number of hours following a first ketamne infusion, consisting of rash and hypertension with no airway interference or swelling. Deemed more likely penicillin allergy. Resolved within hours, no treatment.
Urticaria (Immune system disorders) | 0 (0) | 1 (1) — Pruritis and urticaria developing two days after the first midazolam infusion, other likely contributors identified (laundry detergent). Resolved with oral antihistamine.

LIMITATIONS AND CAVEATS:
Recruitment and randomisation rates in this pilot trial were low, leading to small participant numbers analysed. Due to the potential for breach of confidentiality, limited participant-level information has been reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT02661061/Prot_SAP_000.pdf